CLINICAL TRIAL: NCT01987388
Title: Metabolic Flexibility as a Biomarker of Adaptation to Diet and Exercise Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Rumpler, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HS42
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Intensity Exercise, High Carbohydrate Beverage (Experimental): Study participant consumes a high carbohydrate beverage as part of the day's meals, and performs high intensity exercise (85% of VO2 max), while in the calorimeter.
  Interventions: Other: High Intensity Exercise; Other: High Carbohydrate Beverage
- High Intensity Exercise, High Fat Beverage (Experimental): Study participant consumes a high fat beverage as part of the day's meals, and performs high intensity exercise (85% of VO2 max), while in the calorimeter.
  Interventions: Other: High Intensity Exercise; Other: High Fat Beverage
- Low Intensity Exercise, High Carbohydrate Beverage (Experimental): Study participant consumes a high carbohydrate beverage as part of the day's meals, and performs low intensity exercise (65% of VO2 max), while in the calorimeter.
  Interventions: Other: Low Intensity Exercise; Other: High Carbohydrate Beverage
- Low Intensity Exercise, High Fat Beverage (Experimental): Study participant consumes a high fat beverage as part of the day's meals, and performs low intensity exercise (65% of VO2 max), while in the calorimeter.
  Interventions: Other: Low Intensity Exercise; Other: High Fat Beverage

INTERVENTIONS:
Other: High Intensity Exercise — While in the calorimeter, each subject will complete four bouts of exercise. Each bout is approximately 5 minutes in duration at a predetermined speed and elevation to achieve an intensity of 85% of VO2 max according to their fitness level test described previously. Subjects then sit quietly until either the next meal or the next exercise bout.
  Arms: High Intensity Exercise, High Carbohydrate Beverage; High Intensity Exercise, High Fat Beverage
Other: Low Intensity Exercise — While in the calorimeter, each subject completes one exercise bout approximately 40 minutes in duration, at a predetermined speed and elevation, to achieve an intensity of 65% of VO2 max. Subjects then sit quietly until the next meal.
  Arms: Low Intensity Exercise, High Carbohydrate Beverage; Low Intensity Exercise, High Fat Beverage
Other: High Carbohydrate Beverage — Participants will consume a high carbohydrate beverage (750 g) with the following composition: 2.13 MJ/d, 113g carbohydrate, 4g fat, 6g protein.
  Arms: High Intensity Exercise, High Carbohydrate Beverage; Low Intensity Exercise, High Carbohydrate Beverage
Other: High Fat Beverage — Participants will consume a high fat beverage (750 g) with the following composition: 2.11 MJ/d, 8g carbohydrate, 50g fat, 7g protein.
  Arms: High Intensity Exercise, High Fat Beverage; Low Intensity Exercise, High Fat Beverage

SUMMARY:
The objective is to develop a new metabolic flexibility biomarker, which has application in the study of changes diet and exercise on fuel management in humans. The new biomarker involves the characterization of an individual's metabolic flexibility utilizing room calorimeters rather than the current method, which is based on glucose clamp data. It is hypothesized that this new metabolic flexibility method will be a useful and noninvasive biomarker for measuring adaptation to exercise and diet challenges.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 22 to 35 years at beginning of study

Exclusion Criteria:

* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* History or presence of diabetes, kidney disease, liver disease, certain cancers, gastrointestinal, pancreatic, other metabolic diseases, or malabsorption syndromes.
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (for at least 6 months prior to the start of the study)
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program during the next 10 months
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol
* Inclusion and exclusion criteria have been established to recruit a population of individuals across a wide age-range that has typical digestive process

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Metabolic Flexibility by Room Calorimetry | 24 hours
  Participants will stay in a room calorimeter for 24 hours where oxygen consumed and carbon dioxide produced will be measured. Mathematical approaches will use continuous calorimetry data to generate consistent estimates of the gas exchange rates, and hence accurate "instantaneous" respiratory exchange ratios. This novel approach allows evaluating the instantaneous dynamics of respiratory quotient noninvasively and for many different conditions (e.g., exercise and various nutrient ratios).

SECONDARY OUTCOMES:
Continuous Glucose Monitoring | 24 hours
  Whole-day interstitial glucose profiles will be collected during each calorimeter measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Center, Beltsville, Maryland, United States